CLINICAL TRIAL: NCT00054483
Title: A Phase I Pharmacokinetic Study of PS341 in Patients With Advanced Malignancies and Varying Degrees of Renal Dysfunction for the CTEP-Sponsored Organ Dysfunction Working Group
Brief Title: Bortezomib in Treating Patients With Advanced Cancer and Kidney Dysfunction
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: NCI-2012-02917; CO 02903; CDR0000270687; U01CA062491 (NIH); U01CA069852 (NIH); U01CA062505 (NIH); U01CA062487 (NIH); U01CA069853 (NIH); U01CA062502 (NIH); U01CA099168 (NIH)
Record Dates: First submitted 2003-02-05; First posted 2003-02-06 (Estimated); Last update posted 2013-05-16 (Estimated); Status verified 2013-05

CONDITIONS: Adult Grade III Lymphomatoid Granulomatosis; Adult Nasal Type Extranodal NK/T-cell Lymphoma; Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Nodal Marginal Zone B-cell Lymphoma; Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Diffuse Mixed Cell Lymphoma; Recurrent Adult Diffuse Small Cleaved Cell Lymphoma; Recurrent Adult Grade III Lymphomatoid Granulomatosis; Recurrent Adult Immunoblastic Large Cell Lymphoma; Recurrent Adult Lymphoblastic Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Small Lymphocytic Lymphoma; Refractory Multiple Myeloma; Splenic Marginal Zone Lymphoma; Stage III Multiple Myeloma; Stage IV Adult Burkitt Lymphoma; Stage IV Adult Diffuse Large Cell Lymphoma; Stage IV Adult Diffuse Mixed Cell Lymphoma; Stage IV Adult Diffuse Small Cleaved Cell Lymphoma; Stage IV Adult Immunoblastic Large Cell Lymphoma; Stage IV Adult Lymphoblastic Lymphoma; Stage IV Grade 1 Follicular Lymphoma; Stage IV Grade 2 Follicular Lymphoma; Stage IV Grade 3 Follicular Lymphoma; Stage IV Mantle Cell Lymphoma; Stage IV Marginal Zone Lymphoma; Stage IV Small Lymphocytic Lymphoma; Unspecified Adult Solid Tumor, Protocol Specific; Waldenström Macroglobulinemia
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell; Lymphoma, B-Cell, Marginal Zone; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Leukemia, Lymphocytic, Chronic, B-Cell; Multiple Myeloma; Waldenstrom Macroglobulinemia | interventions — Bortezomib

ARMS (1):
- Treatment (bortezomib) (Experimental): Patients receive bortezomib IV over 3-5 seconds on days 1, 4, 8, and 11. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: bortezomib; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Drug: bortezomib — Given IV
  Other Names: LDP 341; MLN341; VELCADE
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
Phase I trial to study the effectiveness of bortezomib in treating patients who have advanced cancer and kidney dysfunction. Bortezomib may stop the growth of cancer cells by blocking the enzymes necessary for cancer cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To identify the pharmacokinetic and pharmacodynamic profile of PS-341 in patients with advanced malignancy and mild, moderate or severe renal insufficiency.

II. Evaluate the safety, tolerability, and the maximum tolerated dose of PS-341 for patients with varying degrees of renal insufficiency.

OUTLINE: This is a dose-escalation, multicenter study. Patients are stratified according to most recent creatinine clearance (greater than 60 mL/min vs 40-59 mL/min vs 20-39 mL/min vs less than 20 mL/min vs any creatinine clearance and undergoing renal dialysis).

Patients receive bortezomib IV over 3-5 seconds on days 1, 4, 8, and 11. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of bortezomib until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, an additional cohort of up to 12 patients is treated at the MTD.

PROJECTED ACCRUAL: A total of 60-69 patients (at least 12 per stratum) will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Histologic proof of malignancy (including non-Hodgkin's lymphoma and multiple myeloma)
* Patients must have measurable or evaluable disease; patients with reliable tumor markers (as determined by protocol chairman) are eligible for participation
* ANC >= 1000/uL
* PLT >= 50,000/uL
* Total bilirubin =< 1.5 x upper limit of normal (ULN)
* AST =< 2.5 x ULN or AST =< 5 x ULN if liver involvement
* Patients with abnormal kidney function will be allowed and will be grouped accordingly
* Willingness to return to treating institution for follow-up
* Life expectancy >= 12 weeks
* Willingness to provide all biologic specimens as required by the protocol

Exclusion Criteria:

* Known standard therapy for the patient's disease that is potentially curative or definitely capable of extending life expectancy
* ECOG performance status (PS) 3 or 4
* Uncontrolled intercurrent illness including but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Any of the following prior therapies:

  * Chemotherapy ≤ 4 weeks
  * Mitomycin C/nitrosoureas ≤ 6 weeks
  * Immunotherapy ≤ 4 weeks
  * Biologic therapy ≤ 4 weeks
  * Radiation therapy ≤ 2 weeks
  * Radiation to > 50 % of bone marrow (excepting patients who have had total body irradiation incorporated into bone marrow or stem cell transplantation; all other eligibility criteria still apply)
  * PS-341 treatment
* Failure to fully recover from effects of prior chemotherapy regardless of interval since last treatment (excludes renal function)
* New York Heart Association classification III or IV
* Symptomatic CNS metastases; patients who have received definitive treatment for brain metastases (radiation and/or surgery) and are stable for >= 8 weeks are eligible; eligible patients with brain metastases should not be taking enzyme-inducing anticonvulsants and should be receiving stable doses of steroids
* Any of the following:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception (condoms, diaphragm, birth control pills, injections, intrauterine device [IUD], or abstinence, etc.)
  * This study involves an investigational agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown
* Other concurrent chemotherapy, immunotherapy, or radiotherapy
* HIV-positive patients receiving anti-retroviral therapy (HAART); there is a potential for pharmacokinetic interactions
* Concurrent use of other investigational agent (including thalidomide); bisphosphonate therapy (e.g. pamidronate or zoledronate) will not be considered investigational agents for the purpose of trial eligibility
* Pre-existing grade >= 2 neuropathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2003-01; Primary Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics in terms of 20S proteasome activity following bortezomib administration | Days 1 and 8 pre-infusion (of course 1) and 5, 15, 30, and 60 minutes, and 2, 4, 6, 8, 12, and 24 hours post-bortezomib administration
Dose-limiting toxicities of bortezomib graded according to the National Cancer Institute Common Toxicity Criteria (NCI CTC) v2.0 | Up to 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Mulkerin, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Hospital and Clinics, Madison, Wisconsin, United States